CLINICAL TRIAL: NCT03664466
Title: Astaxanthin Effects on Osteoarthritis Associated Pain and Inflammatory Indicators
Acronym: AXE OA PAIN
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Inadequate funding
Sponsor: Saint Luke's Health System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: AXE OA PAIN
Record Dates: First submitted 2018-05-31; First posted 2018-09-10 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-04

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — astaxanthine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Astaxanthin (Experimental): Astaxanthin 12mg twice daily by mouth
  Interventions: Dietary Supplement: astaxanthin
- Placebo (Placebo Comparator): Placebo twice daily by mouth
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: astaxanthin — astaxanthin capsules 12 mg twice daily
  Arms: Astaxanthin
Other: Placebo — placebo capsules twice daily
  Arms: Placebo

SUMMARY:
This study is intended to assess the effects of astaxanthin use on pain, physical function, and inflammation as reflected by Patient-Reported Outcomes Measurement Information System (PROMIS) scores and levels of inflammatory biomarkers in subjects taking astaxanthin. If improvements in pain, function, and/or markers of inflammation could be demonstrated with the use of astaxanthin, this may suggest the potential for astaxanthin to be used in management of knee osteoarthritis (and possibly other forms of osteoarthritis) with less evident toxicity than seen with the presently available standard therapies (e.g. NSAIDS, opioids).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Symptoms of knee pain
* Radiographic evidence of mild to moderate arthritis
* Able to provide written consent on their own behalf

Exclusion Criteria:

* Pregnancy
* Current tobacco use
* Current substance abuse (alcohol or drug)
* Presence of significant cardiovascular, pulmonary, hepatic, or renal disease
* Prior history of knee trauma or surgery
* Gout or pseudogout
* Significant depression or anxiety scores on PHQ-9 and GAD-7, or pre-existing diagnosis of a significant mental health disorder
* Presence of other chronic pain syndromes such as chronic low back or neck pain, fibromyalgia, or complex regional pain syndrome
* Presence of systemic inflammatory conditions such as rheumatoid arthritis, systemic lupus erythematosus, inflammatory bowel disease
* Symptomatic involvement of multiple other joints with osteoarthritis
* Known allergy to fish or astaxanthin
* BMI greater than 35
* Participation in another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-04-29 (Actual); Primary Completion 2022-01-25 (Actual); Study Completion 2022-01-25 (Actual)

PRIMARY OUTCOMES:
Change in PROMIS Numeric Rating Pain Scale | 20 weeks
  Pain improvement in subjects is the primary outcome measure. The Patient Reported Outcomes Measurement Information Systems (PROMIS) Pain Intensity Scale 1a tool will be used. This scale ranges from 0-10, with 0 representing no pain and 10 representing the worst pain imaginable.

SECONDARY OUTCOMES:
Change in PROMIS Pain interference score | 20 weeks
  Reduction in pain interference is a secondary outcome measure. The Patient Reported Outcomes Measurement Information Systems (PROMIS) Pain Interference Short Form 6b will be used as the survey tool for pain interference. This is a set of 6 questions to assess the degree to which pain has interfered with daily activities. There are 5 levels of pain interference from 0 (none at all) to 5 (very much or always). The higher the score, the greater the pain interference.
Change in PROMIS Physical function score | 20 weeks
  Improvement in physical function is a secondary outcome measure. The PROMIS Physical Function Short Form 6b will be used as the survey tool for physical limitation. There are 5 levels of limitation to physical function from 0 (without any difficulty) to 5 (unable to do). The higher the score, the greater the limitation
Change in Erythrocyte Sedimentation Rate | 20 weeks
  Change in ESR (mm/hr)
Change in C-reactive protein levels | 20 weeks
  Change in CRP levels (mg/L)
Change in Interleukin-6 levels | 20 weeks
  Change in IL-6 levels (pg/mL)
Change in Cartilage Oligomeric Matrix Protein levels | 20 weeks
  Change in COMP levels (ng/mL)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Elliott, MD, Principal Investigator — St. Luke's Hospital, Kansas City, Missouri
Locations (1):
- Saint Luke's Hospital of Kansas City, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Altman R, Asch E, Bloch D, Bole G, Borenstein D, Brandt K, Christy W, Cooke TD, Greenwald R, Hochberg M, et al. Development of criteria for the classification and reporting of osteoarthritis. Classification of osteoarthritis of the knee. Diagnostic and Therapeutic Criteria Committee of the American Rheumatism Association. Arthritis Rheum. 1986 Aug;29(8):1039-49. doi: 10.1002/art.1780290816. PMID 3741515
- [Background] Sokolove J, Lepus CM. Role of inflammation in the pathogenesis of osteoarthritis: latest findings and interpretations. Ther Adv Musculoskelet Dis. 2013 Apr;5(2):77-94. doi: 10.1177/1759720X12467868. PMID 23641259
- [Background] Cross M, Smith E, Hoy D, Nolte S, Ackerman I, Fransen M, Bridgett L, Williams S, Guillemin F, Hill CL, Laslett LL, Jones G, Cicuttini F, Osborne R, Vos T, Buchbinder R, Woolf A, March L. The global burden of hip and knee osteoarthritis: estimates from the global burden of disease 2010 study. Ann Rheum Dis. 2014 Jul;73(7):1323-30. doi: 10.1136/annrheumdis-2013-204763. Epub 2014 Feb 19. PMID 24553908
- [Background] Centers for Disease Control and Prevention (CDC). Prevalence and most common causes of disability among adults--United States, 2005. MMWR Morb Mortal Wkly Rep. 2009 May 1;58(16):421-6. PMID 19407734
- [Background] Murphy L, Helmick CG. The impact of osteoarthritis in the United States: a population-health perspective. Am J Nurs. 2012 Mar;112(3 Suppl 1):S13-9. doi: 10.1097/01.NAJ.0000412646.80054.21. PMID 22373741
- [Background] Centers for Disease Control and Prevention (CDC). National and state medical expenditures and lost earnings attributable to arthritis and other rheumatic conditions--United States, 2003. MMWR Morb Mortal Wkly Rep. 2007 Jan 12;56(1):4-7. PMID 17218935
- [Background] Hochberg MC. Mortality in osteoarthritis. Clin Exp Rheumatol. 2008 Sep-Oct;26(5 Suppl 51):S120-4. PMID 19026154
- [Background] Coxib and traditional NSAID Trialists' (CNT) Collaboration; Bhala N, Emberson J, Merhi A, Abramson S, Arber N, Baron JA, Bombardier C, Cannon C, Farkouh ME, FitzGerald GA, Goss P, Halls H, Hawk E, Hawkey C, Hennekens C, Hochberg M, Holland LE, Kearney PM, Laine L, Lanas A, Lance P, Laupacis A, Oates J, Patrono C, Schnitzer TJ, Solomon S, Tugwell P, Wilson K, Wittes J, Baigent C. Vascular and upper gastrointestinal effects of non-steroidal anti-inflammatory drugs: meta-analyses of individual participant data from randomised trials. Lancet. 2013 Aug 31;382(9894):769-79. doi: 10.1016/S0140-6736(13)60900-9. Epub 2013 May 30. PMID 23726390
- [Background] National Center for Health Statistics (US). Health, United States, 2014: With Special Feature on Adults Aged 55-64. Hyattsville (MD): National Center for Health Statistics (US); 2015 May. Report No.: 2015-1232. Available from http://www.ncbi.nlm.nih.gov/books/NBK299348/ PMID 26086064
- [Background] CDC. Multiple cause of death data on CDC WONDER. Atlanta, GA: US Department of Health and Human Services, CDC; 2016. http://wonder.cdc.gov/mcd.html
- [Background] Centers for Disease Control and Prevention (CDC). Vital signs: overdoses of prescription opioid pain relievers---United States, 1999--2008. MMWR Morb Mortal Wkly Rep. 2011 Nov 4;60(43):1487-92. PMID 22048730
- [Background] Dowell D, Haegerich TM, Chou R. CDC Guideline for Prescribing Opioids for Chronic Pain - United States, 2016. MMWR Recomm Rep. 2016 Mar 18;65(1):1-49. doi: 10.15585/mmwr.rr6501e1. PMID 26987082
- [Background] Le Graverand-Gastineau MP. Disease modifying osteoarthritis drugs: facing development challenges and choosing molecular targets. Curr Drug Targets. 2010 May;11(5):528-35. doi: 10.2174/138945010791011893. PMID 20199396
- [Background] Astaxanthin as a pigmenter in salmon feed. Chemicals HVF. Hoffman-La Roche Inc., 1987.
- [Background] Higuera-Ciapara I, Felix-Valenzuela L, Goycoolea FM. Astaxanthin: a review of its chemistry and applications. Crit Rev Food Sci Nutr. 2006;46(2):185-96. doi: 10.1080/10408690590957188. PMID 16431409
- [Background] Spiller GA, Dewell A. Safety of an astaxanthin-rich Haematococcus pluvialis algal extract: a randomized clinical trial. J Med Food. 2003 Spring;6(1):51-6. doi: 10.1089/109662003765184741. PMID 12804020
- [Background] Okada Y, Ishikura M, Maoka T. Bioavailability of astaxanthin in Haematococcus algal extract: the effects of timing of diet and smoking habits. Biosci Biotechnol Biochem. 2009 Sep;73(9):1928-32. doi: 10.1271/bbb.90078. Epub 2009 Sep 7. PMID 19734684
- [Background] Mercke Odeberg J, Lignell A, Pettersson A, Hoglund P. Oral bioavailability of the antioxidant astaxanthin in humans is enhanced by incorporation of lipid based formulations. Eur J Pharm Sci. 2003 Jul;19(4):299-304. doi: 10.1016/s0928-0987(03)00135-0. PMID 12885395
- [Background] Yoshida H, Yanai H, Ito K, Tomono Y, Koikeda T, Tsukahara H, Tada N. Administration of natural astaxanthin increases serum HDL-cholesterol and adiponectin in subjects with mild hyperlipidemia. Atherosclerosis. 2010 Apr;209(2):520-3. doi: 10.1016/j.atherosclerosis.2009.10.012. Epub 2009 Oct 14. PMID 19892350
- [Background] Miyawaki H, Takahashi J, Tsukahara H, Takehara I. Effects of astaxanthin on human blood rheology. J Clin Biochem Nutr. 2008 Sep;43(2):69-74. doi: 10.3164/jcbn.2008048. PMID 18818755
- [Background] Iwabayashi M et al., Efficacy and safety of eight-week treatment with astaxanthin in individuals screened for increased oxidative stress burden. Anti-aging medicine. 2009;6(4):15-21.
- [Background] Pashkow FJ, Watumull DG, Campbell CL. Astaxanthin: a novel potential treatment for oxidative stress and inflammation in cardiovascular disease. Am J Cardiol. 2008 May 22;101(10A):58D-68D. doi: 10.1016/j.amjcard.2008.02.010. PMID 18474276
- [Background] Hussein G, Nakagawa T, Goto H, Shimada Y, Matsumoto K, Sankawa U, Watanabe H. Astaxanthin ameliorates features of metabolic syndrome in SHR/NDmcr-cp. Life Sci. 2007 Jan 16;80(6):522-9. doi: 10.1016/j.lfs.2006.09.041. Epub 2006 Oct 12. PMID 17074368
- [Background] Kim KY et al., The effects of astaxanthin supplements on lipid peroxidation and antioxidant status in postmenopausal women. Nutritional Sciences. 2004;7(1):41-46.
- [Background] Lee SJ, Bai SK, Lee KS, Namkoong S, Na HJ, Ha KS, Han JA, Yim SV, Chang K, Kwon YG, Lee SK, Kim YM. Astaxanthin inhibits nitric oxide production and inflammatory gene expression by suppressing I(kappa)B kinase-dependent NF-kappaB activation. Mol Cells. 2003 Aug 31;16(1):97-105. PMID 14503852
- [Background] Lu YP, Liu SY, Sun H, Wu XM, Li JJ, Zhu L. Neuroprotective effect of astaxanthin on H(2)O(2)-induced neurotoxicity in vitro and on focal cerebral ischemia in vivo. Brain Res. 2010 Nov 11;1360:40-8. doi: 10.1016/j.brainres.2010.09.016. Epub 2010 Sep 21. PMID 20846510
- [Background] Hussein G, Goto H, Oda S, Iguchi T, Sankawa U, Matsumoto K, Watanabe H. Antihypertensive potential and mechanism of action of astaxanthin: II. Vascular reactivity and hemorheology in spontaneously hypertensive rats. Biol Pharm Bull. 2005 Jun;28(6):967-71. doi: 10.1248/bpb.28.967. PMID 15930728
- [Background] Lee DH, Kim CS, Lee YJ. Astaxanthin protects against MPTP/MPP+-induced mitochondrial dysfunction and ROS production in vivo and in vitro. Food Chem Toxicol. 2011 Jan;49(1):271-80. doi: 10.1016/j.fct.2010.10.029. Epub 2010 Nov 5. PMID 21056612
- [Background] Haines DD, Varga B, Bak I, Juhasz B, Mahmoud FF, Kalantari H, Gesztelyi R, Lekli I, Czompa A, Tosaki A. Summative interaction between astaxanthin, Ginkgo biloba extract (EGb761) and vitamin C in suppression of respiratory inflammation: a comparison with ibuprofen. Phytother Res. 2011 Jan;25(1):128-36. doi: 10.1002/ptr.3160. PMID 20632299
- [Background] KELLGREN JH, LAWRENCE JS. Radiological assessment of osteo-arthrosis. Ann Rheum Dis. 1957 Dec;16(4):494-502. doi: 10.1136/ard.16.4.494. No abstract available. PMID 13498604
- [Background] Verma P, Dalal K. Serum cartilage oligomeric matrix protein (COMP) in knee osteoarthritis: a novel diagnostic and prognostic biomarker. J Orthop Res. 2013 Jul;31(7):999-1006. doi: 10.1002/jor.22324. Epub 2013 Feb 19. PMID 23423905
- [Background] Spector TD, Hart DJ, Nandra D, Doyle DV, Mackillop N, Gallimore JR, Pepys MB. Low-level increases in serum C-reactive protein are present in early osteoarthritis of the knee and predict progressive disease. Arthritis Rheum. 1997 Apr;40(4):723-7. doi: 10.1002/art.1780400419. PMID 9125256
- [Background] Tseng S, Reddi AH, Di Cesare PE. Cartilage Oligomeric Matrix Protein (COMP): A Biomarker of Arthritis. Biomark Insights. 2009 Feb 17;4:33-44. doi: 10.4137/bmi.s645. PMID 19652761
- [Background] Attur M, Krasnokutsky-Samuels S, Samuels J, Abramson SB. Prognostic biomarkers in osteoarthritis. Curr Opin Rheumatol. 2013 Jan;25(1):136-44. doi: 10.1097/BOR.0b013e32835a9381. PMID 23169101
- [Background] Crane EH. Highlights of the 2011 Drug Abuse Warning Network (DAWN) Findings on Drug-Related Emergency Department Visits. 2013 Feb 22. In: The CBHSQ Report. Rockville (MD): Substance Abuse and Mental Health Services Administration (US); 2013-. Available from http://www.ncbi.nlm.nih.gov/books/NBK384680/ PMID 27631059
- [Background] Bruyere O, Honore A, Ethgen O, Rovati LC, Giacovelli G, Henrotin YE, Seidel L, Reginster JY. Correlation between radiographic severity of knee osteoarthritis and future disease progression. Results from a 3-year prospective, placebo-controlled study evaluating the effect of glucosamine sulfate. Osteoarthritis Cartilage. 2003 Jan;11(1):1-5. doi: 10.1053/joca.2002.0848. PMID 12505481
- [Background] Jin X, Jones G, Cicuttini F, Wluka A, Zhu Z, Han W, Antony B, Wang X, Winzenberg T, Blizzard L, Ding C. Effect of Vitamin D Supplementation on Tibial Cartilage Volume and Knee Pain Among Patients With Symptomatic Knee Osteoarthritis: A Randomized Clinical Trial. JAMA. 2016 Mar 8;315(10):1005-13. doi: 10.1001/jama.2016.1961. PMID 26954409
- [Background] Geba GP, Weaver AL, Polis AB, Dixon ME, Schnitzer TJ; Vioxx, Acetaminophen, Celecoxib Trial (VACT) Group. Efficacy of rofecoxib, celecoxib, and acetaminophen in osteoarthritis of the knee: a randomized trial. JAMA. 2002 Jan 2;287(1):64-71. doi: 10.1001/jama.287.1.64. PMID 11754710
- [Background] Bellamy N. The WOMAC Knee and Hip Osteoarthritis Indices: development, validation, globalization and influence on the development of the AUSCAN Hand Osteoarthritis Indices. Clin Exp Rheumatol. 2005 Sep-Oct;23(5 Suppl 39):S148-53. PMID 16273799
- [Background] Schumacher HR, Pullman-Mooar S, Gupta SR, Dinnella JE, Kim R, McHugh MP. Randomized double-blind crossover study of the efficacy of a tart cherry juice blend in treatment of osteoarthritis (OA) of the knee. Osteoarthritis Cartilage. 2013 Aug;21(8):1035-41. doi: 10.1016/j.joca.2013.05.009. Epub 2013 May 31. PMID 23727631
- [Background] Pincus T, Koch G, Lei H, Mangal B, Sokka T, Moskowitz R, Wolfe F, Gibofsky A, Simon L, Zlotnick S, Fort JG. Patient Preference for Placebo, Acetaminophen (paracetamol) or Celecoxib Efficacy Studies (PACES): two randomised, double blind, placebo controlled, crossover clinical trials in patients with knee or hip osteoarthritis. Ann Rheum Dis. 2004 Aug;63(8):931-9. doi: 10.1136/ard.2003.020313. Epub 2004 Apr 13. PMID 15082468
- [Background] McConnell S, Kolopack P, Davis AM. The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC): a review of its utility and measurement properties. Arthritis Rheum. 2001 Oct;45(5):453-61. doi: 10.1002/1529-0131(200110)45:53.0.co;2-w. No abstract available. PMID 11642645
- [Background] Augusti PR, Quatrin A, Somacal S, Conterato GM, Sobieski R, Ruviaro AR, Maurer LH, Duarte MM, Roehrs M, Emanuelli T. Astaxanthin prevents changes in the activities of thioredoxin reductase and paraoxonase in hypercholesterolemic rabbits. J Clin Biochem Nutr. 2012 Jul;51(1):42-9. doi: 10.3164/jcbn.11-74. Epub 2012 Jun 8. PMID 22798712
- [Background] Choi HD, Kim JH, Chang MJ, Kyu-Youn Y, Shin WG. Effects of astaxanthin on oxidative stress in overweight and obese adults. Phytother Res. 2011 Dec;25(12):1813-8. doi: 10.1002/ptr.3494. Epub 2011 Apr 8. PMID 21480416
- [Background] Scanzello CR, Goldring SR. The role of synovitis in osteoarthritis pathogenesis. Bone. 2012 Aug;51(2):249-57. doi: 10.1016/j.bone.2012.02.012. Epub 2012 Feb 22. PMID 22387238
- [Background] Miller RE, Miller RJ, Malfait AM. Osteoarthritis joint pain: the cytokine connection. Cytokine. 2014 Dec;70(2):185-93. doi: 10.1016/j.cyto.2014.06.019. Epub 2014 Jul 24. PMID 25066335
- [Background] Goldring MB, Otero M. Inflammation in osteoarthritis. Curr Opin Rheumatol. 2011 Sep;23(5):471-8. doi: 10.1097/BOR.0b013e328349c2b1. PMID 21788902
- [Background] Bondeson J, Blom AB, Wainwright S, Hughes C, Caterson B, van den Berg WB. The role of synovial macrophages and macrophage-produced mediators in driving inflammatory and destructive responses in osteoarthritis. Arthritis Rheum. 2010 Mar;62(3):647-57. doi: 10.1002/art.27290. No abstract available. PMID 20187160
- [Background] Sellam J, Berenbaum F. The role of synovitis in pathophysiology and clinical symptoms of osteoarthritis. Nat Rev Rheumatol. 2010 Nov;6(11):625-35. doi: 10.1038/nrrheum.2010.159. Epub 2010 Oct 5. PMID 20924410
- [Background] Berenbaum F. Osteoarthritis as an inflammatory disease (osteoarthritis is not osteoarthrosis!). Osteoarthritis Cartilage. 2013 Jan;21(1):16-21. doi: 10.1016/j.joca.2012.11.012. Epub 2012 Nov 27. PMID 23194896
- [Background] Malemud CJ. Biologic basis of osteoarthritis: state of the evidence. Curr Opin Rheumatol. 2015 May;27(3):289-94. doi: 10.1097/BOR.0000000000000162. PMID 25784380
- [Background] Rahmati M, Mobasheri A, Mozafari M. Inflammatory mediators in osteoarthritis: A critical review of the state-of-the-art, current prospects, and future challenges. Bone. 2016 Apr;85:81-90. doi: 10.1016/j.bone.2016.01.019. Epub 2016 Jan 23. PMID 26812612
- [Background] Singh S, Shahi NT, Shahi U, Kumar D. Serum Cartilage Oligomeric Matrix Protein (COMP) Estimation: A Tool to Assess Efficacy of Treatment in Knee Osteoarthritis. MOJ Orthopedics & Rheumatology 2014; 1(3): 00017.
- [Background] Stannus O, Jones G, Cicuttini F, Parameswaran V, Quinn S, Burgess J, Ding C. Circulating levels of IL-6 and TNF-alpha are associated with knee radiographic osteoarthritis and knee cartilage loss in older adults. Osteoarthritis Cartilage. 2010 Nov;18(11):1441-7. doi: 10.1016/j.joca.2010.08.016. Epub 2010 Sep 16. PMID 20816981